CLINICAL TRIAL: NCT06519981
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HRS-9231 in Healthy Caucasian Participants
Brief Title: Phase 1 Study of HRS-9231 Safety and Pharmacokinetics in Healthy Caucasians
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HRS-9231-102
Record Dates: First submitted 2024-07-02; First posted 2024-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: MRI

STUDY DESIGN:
Intervention Model Description: Healthy participants are planned to be enrolled in a single ascending dose study. For each cohort, participants will randomly receive HRS-9231/Placebo injection by an intravenous (IV) administration
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-9231 or matching placebo Dose level 1 (Experimental): Dose level 1
  Interventions: Drug: HRS-9231or matching placebo
- HRS-9231 or matching placebo Dose level 2 (Experimental)
  Interventions: Drug: HRS-9231or matching placebo

INTERVENTIONS:
Drug: HRS-9231or matching placebo — HRS-9231 injection or matching placebo will be administered through IV injection.

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled study. The objective of this study is to evaluate the safety, tolerability, and PK profile of HRS-9231 injection following a single dose in healthy Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian participants;
2. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial,
3. Male or female aged between 18 to 45 years of age (inclusive) at the date of signed consent form.
4. Women with body weight of ≥ 45.0 kg, men with body weight ≥ 50.0 kg, body mass Index (BMI) between 18.0 and 32.0 kg/m2

Exclusion Criteria:

1. History or evidence of clinically significant disorders
2. Individuals with a history of drug allergies, specific allergies
3. Severe infections, injuries, or major surgeries as determined by the investigator within 3 months prior to dosing, or plan to do surgeries during the study.
4. Any other circumstances (e.g., not suitable for venous access) or laboratory
5. abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the Study or could preclude the evaluation of the participant's response.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Adverse events | Day 8
  Number of patients with adverse events (AEs) and serious adverse event (SAE)
Vital signs | Day 8
  Number of patients with clinically significant change from baseline in vital signs values
Physical examination | Day 8
  Number of patients with clinically significant change in physical examination
Laboratory | Day 8
  Number of patients with clinically significant change from baseline in laboratory examination
ECG | Day 8
  Number of patients with clinically significant change from baseline in 12-ECG values
Injection site reaction | Day 8
  Number of patients with injection site reaction

SECONDARY OUTCOMES:
Pharmacokinetics PK Cmax | Day 1
  Plasma Pharmacokinetics: Cmax
Pharmacokinetics PK AUC0-t | Day 1
  Plasma Pharmacokinetics: AUC0-t
Pharmacokinetics PK AUC0-inf | Day 1
  Plasma Pharmacokinetics: AUC0-inf
Pharmacokinetics PK Tmax | Day 1
  Plasma Pharmacokinetics: Tmax
Pharmacokinetics PK t1/2 | Day 1
  Plasma Pharmacokinetics: t1/2
Pharmacokinetics PK CL | Day 1
  Plasma Pharmacokinetics: CL
Pharmacokinetics PK Vz | Day 1
  Plasma Pharmacokinetics: Vz
Pharmacokinetics PK MRTlast | Day 1
  Plasma Pharmacokinetics: MRTlast
Pharmacokinetics PK MRTinf | Day 1
  Plasma Pharmacokinetics: MRTinf
Pharmacokinetics PK Ae | Day 3
  Urine Pharmacokinetics: Ae
Pharmacokinetics PK ur | Day 3
  Urine Pharmacokinetics: ur
Pharmacokinetics PK %Ae | Day 3
  Urine Pharmacokinetics: %Ae
Pharmacokinetics PK CLr | Day 3
  Urine Pharmacokinetics: CLr

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical research, Perth, Western Australia, Australia